CLINICAL TRIAL: NCT04569695
Title: A Phase 1, Randomized, Open-label, Parallel-group, Single- and Multiple-dose Study to Characterize Pharmacokinetics, Pharmacodynamics and Safety and Tolerability of JNJ-70033093 (BMS-986177) in Healthy Chinese Adult Subjects
Brief Title: A Study of JNJ-70033093 (BMS-986177) in Healthy Chinese Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CR108806; 70033093THR1003 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2020-09-11; First posted 2020-09-30 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Healthy
MeSH Terms: interventions — milvexian

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Part 1: Cohort A: JNJ-70033093 (Experimental): Participants will receive Dose 1 of JNJ-70033093 once daily (QD) on Day 1 followed by washout period of 4 days and then Dose 1 of JNJ-70033093 QD from Days 5 to 12.
  Interventions: Drug: JNJ-70033093
- Part 1: Cohort B: JNJ-70033093 (Experimental): Participants will receive Dose 1 of JNJ-70033093 twice daily (BID) from Days 1 to 8.
  Interventions: Drug: JNJ-70033093
- Part 1: Cohort C: JNJ-70033093 (Experimental): Participants will receive Dose 2 of JNJ-70033093 BID from Days 1 to 8.
  Interventions: Drug: JNJ-70033093
- Part 2: Cohort D: JNJ-70033093 (Experimental): Participants will receive Dose 3 of JNJ-70033093 QD on Day 1 followed by washout period of 4 days and then Dose 3 of JNJ-70033093 BID from Days 5 to 12 in Cohort D. Dose escalation to Part 2: Cohort D will occur only after the safety and tolerability data of the Part 1 are assessed.
  Interventions: Drug: JNJ-70033093

INTERVENTIONS:
Drug: JNJ-70033093 — JNJ-70033093 capsule will be administered orally as per assigned treatment regimen.
  Other Names: BMS-986177

SUMMARY:
The purpose of the study is to characterize the pharmacokinetics of single and multiple doses of JNJ-70033093 (BMS-986177) in healthy Chinese participants.

ELIGIBILITY:
Inclusion criteria:

* Healthy on the basis of physical examination, medical history, vital signs, Electrocardiogram (ECG), and the results of serum biochemistry, blood coagulation and hematology test and a urinalysis performed at screening. If there are abnormalities, investigator judges the abnormalities or deviations from normal to be not clinically significant. This determination must be recorded in the subject's source documents and initialed by the investigator
* Must sign an Informed consent Form (ICF) indicating that they understand the purpose of, and procedures required for the study and is willing to participate in the study
* If a woman, except for postmenopausal women, must have a negative highly sensitive serum (beta human chorionic gonadotropin [beta hCG]) at screening and urine (beta-hCG) pregnancy test on Day -1
* Contraceptive use by men or women should be consistent with local regulations regarding the use of contraceptive methods for subject participating in clinical studies
* Before randomization, a woman must be either not of childbearing potential; of childbearing potential and practicing a highly effective method of contraception and agrees to remain on a highly effective method throughout the study and for at least 34 days after the last dose of study drug; women must have no history of excessive menstrual bleeding or hemorrhage following pregnancy delivery

Exclusion criteria:

* If a woman, pregnant, breast-feeding or planning to become pregnant during the study
* Participants with current hepatitis B infection (confirmed by hepatitis B surface antigen [HBsAg]), or hepatitis C infection (confirmed by hepatitis C virus [HCV] antibody), or human immunodeficiency virus type-1 (HIV-1) or HIV-2 infection at study screening
* History of, or a reason to believe a subject has a history of, drug or alcohol abuse within the past 1 year, which in the Investigator's opinion would compromise subject's safety and/or compliance with the study procedures
* History of any significant drug allergy (such as anaphylaxis or hepatotoxicity) and known allergy to the study drug or any of the excipients of the formulation
* Preplanned surgery or procedures that would interfere with the conduct of the study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2021-03-08 (Actual); Primary Completion 2021-12-04 (Actual); Study Completion 2021-12-16 (Actual)

PRIMARY OUTCOMES:
Cohort A and D: Plasma Concentration of JNJ-70033093 After Single Dose Administration | Up to Day 15 (Cohort A and D) and up to Day 11 (Cohort C and B)
  Plasma concentration of JNJ-70033093 after single dose administration will be analyzed.
Cohort A, B, C and D: Plasma Concentration of JNJ-70033093 After Multiple Dose Administration | Up to Day 15 (Cohort A and D) and up to Day 11 (Cohort C and B)
  Observed plasma concentration of JNJ-70033093 after multiple dose administration will be analyzed.

SECONDARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | Up to 54 Days
  Number of participants who experience at least 1 occurrence of each treatment emergent adverse event (TEAE) will be assessed.
Number of Participants with Clinical Laboratory Abnormalities | Up to 54 Days
  Number of participants with clinical laboratories (such as Hematology, Coagulation, Serum chemistry and urinalysis) abnormalities will be assessed.
Number of Participants with Vital Signs Abnormalities | Up to 54 Days
  Number of participants with vital sign abnormalities (such as, blood pressure, pulse, respiratory rate, and temperature) will be assessed.
Change From Baseline in Activated Partial Thromboplastin Time (aPTT) | Up to Day 15 (Cohort A and D) and up to Day 11 (Cohort C and B)
  Activated partial thromboplastin time measures the time to clot formation via the intrinsic (contact) and common pathways, and is dependent on activation of contact factors (such as FXI).
Percentage Change From Baseline in FXI Clotting Activity | Up to Day 15 (Cohort A and D) and up to Day 11 (Cohort C and B)
  Percentage change from baseline in FXI clotting activity will be measured using a modified aPTT assay.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- West China Hospital Si Chuan University, Chengdu, China

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency